CLINICAL TRIAL: NCT01354002
Title: TBANK: Protocol for Collecting, Banking and Distributing Human Tissue Samples: St. Jude Children's Research Hospital Tissue Resources Core Facility
Brief Title: Protocol for Collecting, Banking and Distributing Human Tissue Samples: St. Jude Children's Research Hospital Tissue Resources Core Facility
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TBANK
Record Dates: First submitted 2011-05-09; First posted 2011-05-16 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Normal and Diseased Tissue and Body Fluids Samples
Keywords: human biological samples; tissue banking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected and processed from patients include any tumor or non-tumor sample, including blood, ascites, pleural effusion, bone marrow, solid tumors, brain tumors, tissue uninvolved by tumor, cerebrospinal fluid, and urine samples. Non-tumor samples are also collected and processed from patients' relatives and controls. Samples are processed under sterile conditions whenever possible, and tumor cells and tissues are cryopreserved viable. Cellular subfractions are also isolated including DNA, RNA, and protein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Protocol Participants: All participants enrolled on protocols

SUMMARY:
The aims of this protocol are: to collect and store diseased and normal tissue and body fluid samples from new and returning patients at St. Jude Children's Research Hospital (SJCRH), affiliated sites and collaborating institutions; to collect and store samples from relatives of SJCRH patients; to collect and store retrospective and prospective pertinent corresponding clinical and laboratory data on disease characterization, treatment, and outcome; and to serve as a source of human biological samples and corresponding laboratory and clinical data.

DETAILED DESCRIPTION:
There is no study design for this protocol. Samples obtained under IRB/IEC-approved protocols that clearly permit storage of patient material at SJCRH will be banked, provided proof of informed consent is available. Such samples will be tagged accordingly and will be only released to fulfill the aim(s) of the protocol under which they were obtained, or to investigators that apply to the St. Jude Children's Research Hospital Tissue Resources Committee to use the samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients (and their relatives) and control populations treated or studied at SJCRH and SJCRH affiliates and collaborating sites that have IRB approval for TBANK with malignant and non-malignant conditions.
* Patients from institutions that do not have Institutional Review Board (IRB) approval for TBANK, and at which a banking mechanism may not be established, who provide samples for research at St. Jude and from whom consent for TBANK is obtained by the TBANK principal investigator (PI).
* Samples from employees of St. Jude Children's Research Hospital (SJCRH) collected for public health surveillance studies (e.g. SJTRC-NCT04362995) provided the employees have consented to participate in the specific IRB-approved studies.

Exclusion Criteria:

* Patients from institutions that do not have IRB approval for TBANK, and who have not provided consent for TBANK, or patients not enrolled on SJCRH protocols that incorporate consent for tumor banking.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients, their relatives, and control populations treated at St. Jude Children's Research Hospital (SJCRH), collaborating sites and affiliates.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2009-09-01 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Collecting, processing and archiving human tissue | Samples will be stored indefinitely.
  Human tissue and body fluids will be collected for use in research; The processing of samples helps to reduce duplication of technical effort, equipment, supplies, and laboratory space by investigators requiring human tissues for research

CONTACTS AND LOCATIONS:
Overall Officials: Charles Mullighan, MBBS, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (14):
- United States (14):
  - St. Jude Clinic at Huntsville Hospital for Women & Children, Huntsville, Alabama
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital and Health Center, San Diego, California
  - Children's Hospital of Illinois at OSF-Saint Francis Medical Center, Peoria, Illinois
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mercy Children's Hospital - Springfield, Springfield, Missouri
  - St. Jude Affiliate Clinic at Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - St. Jude Affiliate Clinic at Saint Francis Children's Hospital, Tulsa, Oklahoma
  - Johnson City Medical Center, Johnson City, Tennessee
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Derived] Maciaszek JL, Oak N, Chen W, Hamilton KV, McGee RB, Nuccio R, Mostafavi R, Hines-Dowell S, Harrison L, Taylor L, Gerhardt EL, Ouma A, Edmonson MN, Patel A, Nakitandwe J, Pappo AS, Azzato EM, Shurtleff SA, Ellison DW, Downing JR, Hudson MM, Robison LL, Santana V, Newman S, Zhang J, Wang Z, Wu G, Nichols KE, Kesserwan CA. Enrichment of heterozygous germline RECQL4 loss-of-function variants in pediatric osteosarcoma. Cold Spring Harb Mol Case Stud. 2019 Oct 23;5(5):a004218. doi: 10.1101/mcs.a004218. Print 2019 Oct. PMID 31604778
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols